CLINICAL TRIAL: NCT06430333
Title: Sleep to Reduce Incident Depression Effectively in Peripartum
Acronym: STRIDE P
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, David Kalmbach, Associate Scientist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STRIDE P
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Insomnia; Depression
Keywords: pregnancy; postpartum; sleep; worry; rumination
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Rumination Syndrome | interventions — Sleep

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perinatal Understanding of Mindful Awareness for Sleep (PUMAS) (Experimental): PUMAS is a clinician-administered psychotherapy intervention for prenatal insomnia that includes six weekly 60-minute sessions in an individual format. PUMAS combines behavioral sleep strategies with mindfulness exercises and tailors all components to pregnancy to improve sleep quality. PUMAS will be delivered via telemedicine video.
  Interventions: Behavioral: Perinatal Understanding of Mindful Awareness for Sleep (PUMAS)
- Treatment-as-usual (TAU) (Active Comparator): TAU reflects real-world care where patients and their providers make their own treatment decisions for treating prenatal insomnia. Common TAU options include over-the-counter sleep aids, sleep hygiene education, melatonin, and cognitive-behavioral therapy for insomnia. The TAU group will be well-characterized (i.e., the investigators will monitor interventions administered by the usual care providers and collect information on dosage, frequency, duration, adherence) to best describe treatment options sought and completed in the real world.
  Interventions: Other: Treatment-as-usual (TAU)

INTERVENTIONS:
Behavioral: Perinatal Understanding of Mindful Awareness for Sleep (PUMAS) — Mindfulness-based sleep program for pregnant women.
  Arms: Perinatal Understanding of Mindful Awareness for Sleep (PUMAS)
Other: Treatment-as-usual (TAU) — Usual practices from real-world care experiences.
  Other Names: Usual care practice
  Arms: Treatment-as-usual (TAU)

SUMMARY:
Perinatal depression (PND) is the most common complication in pregnancy and postpartum, which increases risk for adverse perinatal outcomes such as preterm birth, maternal suicidal thoughts, and impaired mother-infant bonding. Insomnia often precedes PND cases and may serve as an entry point for interventions preventing PND. The proposed project is a large-scale clinical trial to test the effectiveness of a mindfulness-based sleep program designed for pregnant women to improve sleep and alleviate cognitive arousal to reduce risk for PND across pregnancy and postpartum.

DETAILED DESCRIPTION:
Perinatal depression (PND) affects nearly 20% of pregnant and postpartum women, with estimates soaring above 30% during the COVID-19 pandemic. Prospective data show insomnia often precedes PND incidence and relapse cases by more than doubling risk for major depression. This is highly relevant to a large segment of the pregnant population as ~20% of women meet diagnostic criteria for insomnia disorder by the end of pregnancy. Fortunately, insomnia is a modifiable risk factor for PND, and insomnia may serve as an entry point to prevent PND incidence and relapse. The investigators have identified cognitive arousal as a promising candidate factor for alleviating insomnia and preventing depression via insomnia therapy. Indeed, undertreatment of cognitive arousal in pregnancy is associated with insomnia non-remission and continued depression after therapy. Moreover, patient stakeholders identify 'calming a busy mind at night' as a critical target for improving sleep during pregnancy. In effort to enhance alleviation of cognitive arousal to optimize clinical outcomes, the investigators developed Perinatal Understanding of Mindful Awareness for Sleep (PUMAS). PUMAS places behavioral sleep strategies within a mindfulness intervention framework to develop an insomnia therapy specifically for pregnant women: RCT data show that PUMAS yields large effects on insomnia, depression, and cognitive arousal.

This study is a hybrid effectiveness-implementation RCT of 500 women with DSM-5 insomnia disorder (without PND) who are randomized to PUMAS or treatment-as-usual. The investigators will evaluate the effectiveness of PUMAS for alleviating insomnia and preventing PND across pregnancy and the first postpartum year. The investigators will also evaluate whether PUMAS engages a key candidate mechanism (high cognitive arousal) that is operative for addressing these clinical outcomes in the effectiveness context.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy, gestational week 14-31 at screening.
2. DSM-5 Insomnia Disorder (≥1 month duration).
3. Insomnia Severity Index (ISI) score ≥ 11.
4. Edinburgh Postnatal Depression Scale score<13 at screening.
5. No current DSM-5 Major Depression.
6. Reliable internet access for treatment and assessments.
7. Not currently engaged in therapy for major depression or insomnia disorder.
8. Age 18 years or older.

Exclusion Criteria:

1. High risk pregnancy (pre-eclampsia, placenta previa w/ hemorrhage, other conditions deemed serious risk to mother or fetus; hypertension and diabetes are allowed).
2. Active suicidal intent.
3. Night or rotating shift work, anticipated travel across time 3 or more time zones in the 2 months after baseline screening.
4. Untreated RLS (treated RLS is OK).
5. Excessive daytime sleepiness; Epworth Sleepiness Scale>15.
6. Uncontrolled sleep or mental disorder inappropriate or unsafe for sleep restriction (narcolepsy, bipolar, epilepsy, etc.).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Comparative effectiveness between PUMAS and standard care on changes in insomnia symptoms. | The investigators will examine change in ISI from Pretreatment Baseline to Posttreatment (8 weeks after baseline), and monthly for 1 year after childbirth..
  The Insomnia Severity Index is a commonly used self-report measure of insomnia symptoms that has been validated in peripartum. ISI scores range from 0 to 28 with higher scores indicating greater insomnia severity.
Comparative effectiveness of PUMAS and standard care on prevention of perinatal depression. | The investigators will examine onset of perinatal depression (EPDS scores 13 or higher) at posttreatment (8 weeks after baseline) and assessed monthly for 1 year after childbirth.
  The Edinburgh Postnatal Depression Scale (EDPS) is the most widely use depression measure in pregnancy and postpartum. EPDS scores range from 0 to 30 with higher scores indicating greater depression severity.

SECONDARY OUTCOMES:
Comparative effectiveness between PUMAS and standard care on nocturnal cognitive arousal symptoms. | The investigators will examine changes in PSASC from Pretreatment baseline to Posttreatment (8 weeks later).
  The Pre-Sleep Arousal Scale's Cognitive factor (PSASC) is a self-report measure of nocturnal cognitive arousal that has been validated in peripartum. PSASC scores range 8 to 40 with higher scores indicating greater nocturnal cognitive arousal.

CONTACTS AND LOCATIONS:
Overall Officials: David A Kalmbach, PhD, Principal Investigator — Henry Ford Health
Locations (1):
- Henry Ford Medical Center, Novi, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
N/A - The investigators do not plan to share individual participant data to other researchers.